CLINICAL TRIAL: NCT00840489
Title: Phase II Trial of Long-term Monotherapy With Ribavirin Against Colchicine on Progression of Chronic Hepatitis C With Advanced Fibrosis in Patients With Non-response to Standard Antiviral Therapy
Brief Title: Efficacy of Long-term Ribavirin in Non-responders With Chronic Hepatitis C and Advanced Fibrosis
Acronym: RIBACIR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary analysis
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Agustin Albillos, Professor of Medicine, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIBACIR-1
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; Colchicine; colchimax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ribavirin (Experimental): Ribavirin 1000-1200 mg qd
  Interventions: Drug: Ribavirin
- Colchicine (Active Comparator): Colchicine 0.5 mg bd
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Ribavirin — Ribavirin 1000-1200 mg qd for 24 weeks
  Other Names: Rebetol
  Arms: Ribavirin
Drug: Colchicine — Colchicine 0.5 mg bd for 24 weeks
  Other Names: Colchimax
  Arms: Colchicine

SUMMARY:
The rate of sustained virological response to a course of standard antiviral therapy (peg-interferon plus ribavirin) of patients with chronic hepatitis C infected by genotype 1 with advanced fibrosis (>F2) is rather low. Monotherapy with ribavirin reduces ALT levels and necroinflammatory liver activity in up to a half of non-responders to standard antiviral therapy, but without changes in liver fibrosis or viremia. Such a beneficial effect seems to be mainly due to the immunomodulatory effect of ribavirin. Portal pressure, as measured by HVPG, lowers in patients with chronic hepatitis C and advanced fibrosis with end-of-treatment response to peg-interferon plus ribavirin. Portal pressure reduction in this setting relates to a reduction of the necroinflammatory liver activity, but not with fibrosis amelioration. We hypothesize that monotherapy with ribavirin reduces portal pressure in hepatitis C patients with advanced fibrosis by means of its immunomodulatory and anti-inflammatory effects, and could constitute an alternative to non-responders to standard antiviral treatment. Portal pressure measurement has become a validated surrogate outcome measure in chronic liver disease, since decreasing portal pressure has shown consistent improvement in survival and clinical outcomes, such as complications of portal hypertension. The primary aim of this study is to investigate whether ribavirin monotherapy slows the progression of advanced chronic liver disease by hepatitis C as assessed by a reduction in HVPG.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA in serum
* AST/ALT greater than the upper limit of normal range
* HVPG >5 mm Hg
* Non-response or contraindication to a standard course of antiviral therapy

Exclusion Criteria:

* Active alcoholism
* HIV infection
* Serum creatinine >1.2 mg/dl, hemoglobin <11 g/dl, hemolysis, symptomatic ischemic heart disease or cerebrovascular disease
* Decompensated chronic liver disease
* Pregnancy
* Hypersensitivity to the drugs of the study
* Severe concomitant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hepatic disease progression defined by a difference of >2 mmHg in the hepatic venous gradient between the basal values and the end of treatment values in both groups | 24 weeks

SECONDARY OUTCOMES:
Decrease in the necroinflammatory activity and in the progression of fibrosis. Normalization of ALT levels. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Albillos, MD, Principal Investigator — Hospital Universitario Ramón y Cajal; José Luis Calleja, MD, Study Director — Hospital Universitario Puerta de Hierro Majadahonda; Rafael Bañares, MD, Study Director — Hospital General Universitario Gregorio Marañón
Locations (3):
- Spain (3):
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Madrid, Madrid